CLINICAL TRIAL: NCT00369447
Title: A Phase I-II Clinical Study of Nimotuzumab (TheraCIM h-R3) in Combination With External Radiotherapy in Stage IIB, III and IV NSCLC
Brief Title: A Study of Nimotuzumab in Combination With External Radiotherapy in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was closed due to slow accrual.
Sponsor: YM BioSciences (Industry)
Collaborators: CIMYM BioSciences (Other)
Responsible Party: Wendy Chapman, Vice President, Clinical Operations, YM BioSciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YMB1000-010
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Non small cell lung cancer; NSCLC; Nimotuzumab; TheraCIM; h-R3; YM BioSciences; Radiation; Non small cell lung cancer, Stage IIb, III and IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 200 mg dose
  Interventions: Procedure: External radiotherapy; Biological: nimotuzumab
- 2 (Placebo Comparator)
  Interventions: Procedure: External radiotherapy; Biological: nimotuzumab

INTERVENTIONS:
Procedure: External radiotherapy — Radiotherapy for first 2 weeks, 10 daily fractions of 30Gy 2 additional fractions to be added if desirable
Biological: nimotuzumab — weekly dose until disease progression

SUMMARY:
This is a Phase I-II study designed to investigate nimotuzumab (TheraCIM h-R3) in combination with external radiation in patients with non-small cell lung cancer. The purpose of the Phase I portion of the study is to evaluate the safety and feasibility of the administration of nimotuzumab with palliative radiation in patients who are unsuitable for radical therapy and to select the optimal dose for the Phase II component of the study. The primary objective for the Phase II portion of the study is to examine the efficacy of this combination treatment.

The Phase I component of this study has been completed. The Phase II is now closed to recruitment.

DETAILED DESCRIPTION:
This is a randomized, double blind, multicenter Phase II study with Phase I lead-in. Patients enrolled in this study will receive external radiotherapy with or without nimotuzumab (TheraCIM h-R3). The objective of the Phase I component of the study is to evaluate the safety and feasibility of the administration of nimotuzumab with palliative radiation in patients who are unsuitable for radical therapy (curative intent chemoradiation) and to select the optimal biologically effective dose (BED) for Phase II component of the study. In the Phase II component, overall survival, local and systemic response rates and quality of life will be evaluated inpatients treated with nimotuzumab in combination with palliative radiation vs. radiation alone.

The Phase I component of this study has been completed. The Phase II is now closed to recruitment.

ELIGIBILITY:
1. Patients must have histologically or cytologically confirmed non-small cell lung cancer.
2. Patients must be suitable for palliative radiation therapy as per institutional standards.
3. Stage IIB, III or IV (patients off steroids with treated, stable brain metastases are eligible).
4. Patients may be symptomatic or asymptomatic from disease
5. Age >18 years
6. ECOG 0-1-2
7. Patients who received previous chemotherapy are allowed
8. Haemoglobin >9g/dL (blood transfusion to increase Hb level is acceptable)
9. Stage II/III patients must be considered unsuitable for radical (standard full dose curative intent) chemoradiation in the opinion of either the radiotherapist or medical oncologist.
10. Patients must have measurable disease in the planned radiation field.
11. Women of child-bearing potential and men must agree to use adequate contraception.
12. Ability to understand and the willingness to sign a written informed consent document

Exclusion criteria - Phase I and Phase II:

1. Patients receiving any other investigational agents
2. Previous treatment with anti-EGF-R drug(s)
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to nimotuzumab or other agents used in study.
4. Prior thoracic radiotherapy for this condition
5. Prior chemotherapy within 4 weeks of enrolment
6. Lesions not suitable for radiotherapy
7. Patients with known sero positive HIV
8. Patients with uncontrolled hypercalcemia
9. Patients with progressive or untreated brain metastases or treated brain metastases but unable to discontinue steroids
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, severe cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator
11. Pregnant or breast-feeding women
12. Any concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix; patients with other prior malignancies are eligible providing prior malignancy cannot be clinically confused with the diagnosis of NSCLC in the opinion of the treating oncologist; in particular, there should be no evidence of current disease activity with respect to the prior malignancy
13. Life expectancy of less than 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Phase II: Overall survival | Every 8 weeks until disease progression

SECONDARY OUTCOMES:
Phase I: Biologically effective dose | 2.5 Years
Phase II: Overall response rate | Every 8 weeks until disease progression
Local response rate | Every 8 weeks until disease progression
Overall clinical benefit | Every 8 weeks until disease progression
Local clinical benefit | Every 8 weeks until disease progression
Time to progression | Every 8 weeks until disease progression
Time to local progression | Every 8 weeks until disease progression
Progression-free survival | 1 year
Phase II: Quality of life | At week 4, week 8, every 2 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Gwyn Bebb, MD, Principal Investigator — Tom Baker Cancer Center; Anthony Brade, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (13):
- Florida Cancer Institute - New Hope, New Port Richey, Florida, United States
- Canada (11):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - London Regional Cancer Center, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunderbay Regional hospital Center, Thunderbay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de L'Universite de Montreal - Hôpital Notre Dame, Montreal, Quebec
  - Segal Cancer Center - Jewish General Hospital, Montreal, Quebec
  - Hotel Dieu Hospital, Québec, Quebec
- National Cancer Center Singapore, Singapore, Singapore